CLINICAL TRIAL: NCT00814671
Title: A Phase 2 Randomized, Open-label Trial of Daily Rifapentine 450mg or 600mg in Place of Rifampicin 600mg for Intensive Phase Treatment of Smear-positive Pulmonary Tuberculosis
Brief Title: Study of Daily Rifapentine for Pulmonary Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Cape Town Lung Institute (Other); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00019095
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Results first posted 2016-09-28 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Pharmacokinetics
MeSH Terms: conditions — Tuberculosis | interventions — rifapentine; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RPT450 (Experimental): Rifapentine 450mg daily
  Interventions: Drug: Rifapentine 450
- RIF 600 (Active Comparator): Rifampin 600mg daily
  Interventions: Drug: Rifampin
- RPT 600 (Experimental): Rifapentine 600mg daily
  Interventions: Drug: Rifapentine 600

INTERVENTIONS:
Drug: Rifapentine 450 — rifapentine 450 mg
  Other Names: Priftin
  Arms: RPT450
Drug: Rifapentine 600 — rifapentine 600 mg
  Other Names: Priftin
  Arms: RPT 600
Drug: Rifampin — rifampin 600 mg
  Other Names: Rifampacin
  Arms: RIF 600

SUMMARY:
The goal of this Phase 2 study is to determine the microbiological activity and safety of rifapentine when given as a component of multidrug intensive phase treatment of smear-positive pulmonary tuberculosis (TB).

Funding Source- FDA Office of Orphan Products Development (OOPD)

DETAILED DESCRIPTION:
Prospective phase II, open-label, single center study in which each experimental rifapentine regimen is evaluated using a two-stage design. Adults (HIV-negative, or HIV-positive with CD4 > 200 cells/cu mm) suspected to have pulmonary tuberculosis who meet eligibility criteria will be randomized to receive one of three intensive phase regimens. Intensive phase regimens will consist of once daily isoniazid, pyrazinamide, and ethambutol, plus one of the following: rifampin 600 mg once daily OR rifapentine 450 mg once daily OR rifapentine 600 mg once daily. Randomization will be stratified by presence/absence of cavitation on baseline chest radiograph. In Stage 1, 15 subjects will be randomized to each arm, following which there will be an enrollment pause for efficacy and safety assessment. Any rifapentine regimen for which fewer than 6 of 11 evaluable participants have week 8 culture conversion will be discarded.

Stage 2 will randomize subjects into the remaining "accepted arms" with a maximum of 36 additional subjects per arm.

All subjects will continue TB treatment with a conventional continuation phase treatment.

Study Site

Study subjects will be recruited from the University of Cape Town inpatient wards and outpatient clinics.

Estimated Study Duration

It is estimated that 18 months will be required for recruitment and enrollment of study subjects. The estimated duration of participation for each study subject is 18 months, including 2 months of experimental intensive phase TB treatment, 4 months of non-experimental conventional continuation phase TB treatment, and an additional 12 months for follow-up for TB relapse.

Study Management

Study subjects will have study visits on days 0, 7, 14, 21, 28, 35, 42, 49, and 56 for sputum collection and adverse event assessment. Safety laboratory monitoring will be performed on days 14, 28, 42, and 56 and will consist of complete blood count, serum alanine aminotransferase, serum total bilirubin, and serum creatinine. Steady state pharmacokinetic analysis will be performed on approximately day 28. Subjects will have additional study visits at week 10 and at months 4, 6, 12, and 18.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected pulmonary tuberculosis with acid-fast bacilli in a stained smear of expectorated sputum. Patients having extra-pulmonary manifestations of tuberculosis, in addition to smear-positive pulmonary disease, are eligible for enrollment.
2. No prior history of tuberculosis disease or tuberculosis treatment
3. No treatment with fluoroquinolones in the 2 months preceding initiation of study drugs.
4. Age > 18 years
5. Weight ≥ 50 kg and ≤ 80 kg
6. Karnofsky score of at least 60 (requires occasional assistance but is able to care for most of his/her needs; see Appendix)
7. Signed informed consent
8. Ability to adhere with study follow-up
9. Women with child-bearing potential must agree to practice an adequate (barrier) method of birth control or to abstain from heterosexual intercourse during study therapy.
10. HIV negative, or HIV-positive with CD4 > 200 cells/cu mm
11. Laboratory parameters done at, or 14 days prior to, screening (with results available for review by study personnel):

    * Serum alanine aminotransferase (ALT) activity ≤ 2 times the upper limit of normal
    * Serum total bilirubin level ≤ 2 times the upper limit of normal
    * Serum creatinine level less than or equal to the upper limit of normal
    * Hemoglobin level of at least 7.0 g/dL
    * Platelet count of at least 100,000/mm3
    * Negative pregnancy test (women of childbearing potential)

Exclusion Criteria:

1. Pregnant or breast-feeding
2. Known intolerance or allergy to any of the study drugs
3. Concomitant disorders or conditions for which isoniazid (INH), rifamycins, pyrazinamide (PZA), or ethambutol (EMB) are contraindicated. These include severe hepatic damage, acute liver disease of any cause, and acute uncontrolled gouty arthritis.
4. Current or planned therapy, during the intensive phase of TB therapy with cyclosporine or tacrolimus, or HIV antiretroviral (ARV) therapy, which have unacceptable interactions with rifamycins.
5. Any medical or psychosocial condition, which, in the view of the study investigator, makes study participation inadvisable.
6. Pulmonary silicosis
7. Central nervous system TB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2010-04; Primary Completion 2013-06 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Dorman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Universiy of Cape Town Lung Institute, Cape Town, Western Cape, South Africa

REFERENCES:
- [Result] Rosenthal IM, Williams K, Tyagi S, Peloquin CA, Vernon AA, Bishai WR, Grosset JH, Nuermberger EL. Potent twice-weekly rifapentine-containing regimens in murine tuberculosis. Am J Respir Crit Care Med. 2006 Jul 1;174(1):94-101. doi: 10.1164/rccm.200602-280OC. Epub 2006 Mar 30. PMID 16574936
- [Result] Rosenthal IM, Williams K, Tyagi S, Vernon AA, Peloquin CA, Bishai WR, Grosset JH, Nuermberger EL. Weekly moxifloxacin and rifapentine is more active than the denver regimen in murine tuberculosis. Am J Respir Crit Care Med. 2005 Dec 1;172(11):1457-62. doi: 10.1164/rccm.200507-1072OC. Epub 2005 Sep 1. PMID 16141439

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 192 individuals assessed for eligibility, 39 excluded, 153 randomized.
Groups:
- RPT450: Rifapentine 450mg daily
  Rifapentine: rifapentine 450 mg + isoniazid + pyrazinamide + ethambutol once a day, seven days a week for 8 weeks
  Rifapentine: rifapentine 600 mg + isoniazid + pyrazinamide + ethambutol once a day, seven days a week for 8 weeks
- RIF 600: Rifampin 600mg daily
  Rifampin: rifampin 600 mg + isoniazid + pyrazinamide + ethambutol once a day, seven days a week for 8 weeks
- RPT 600: Rifapentine 600mg daily
  Rifapentine: rifapentine 450 mg + isoniazid + pyrazinamide + ethambutol once a day, seven days a week for 8 weeks
  Rifapentine: rifapentine 600 mg + isoniazid + pyrazinamide + ethambutol once a day, seven days a week for 8 weeks
Period: Overall Study
Arm/Group | RPT450 | RIF 600 | RPT 600
Started | 54 | 48 | 51
Completed | 47 | 44 | 49
Not Completed | 7 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RPT450 | RIF 600 | RPT 600 | Total
Number analyzed (Participants) | 54 | 48 | 51 | 153
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [23 to 39] | 30 [25 to 36] | 29 [24 to 38] | 29 [24 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 11 | 37
  Male | 41 | 35 | 40 | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 54 | 48 | 51 | 153
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 54 | 48 | 51 | 153

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Negative Lowenstein Jensen Cultures at Week 8
Time Frame: 8 weeks
Population: per protocol
Measure: Number; unit: percentage of participants w/LJ cx con
Arm/Group | RPT450 | RIF 600 | RPT 600
Number analyzed (Participants) | 41 | 36 | 45
percentage of participants w/LJ cx con | 85 | 94 | 96

2. Primary Outcome: Tolerability
Description: percentage of participants discontinuing assigned treatment
Time Frame: 10 weeks
Population: safety analysis population
Measure: Number; unit: percentage of participants
Arm/Group | RPT450 | RIF 600 | RPT 600
Number analyzed (Participants) | 54 | 48 | 51
percentage of participants | 2.0 | 8.3 | 2.0

3. Secondary Outcome: Time to Stable Culture Conversion on Solid Medium
Description: Time to stable culture conversion (in days) on Lowenstein Jensen solid medium
Time Frame: 12 weeks
Population: Data was not collected on some participants due to loss to follow up
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- RPT450: Rifapentine 450mg daily
  Rifapentine 450: rifapentine 450 mg + isoniazid + pyrazinamide + ethambutol once a day, seven days a week for 8 weeks
- RPT 600: Rifapentine 600mg daily
  Rifapentine 600: rifapentine 600 mg + isoniazid + pyrazinamide + ethambutol once a day, seven days a week for 8 weeks
Arm/Group | RPT450 | RIF 600 | RPT 600
Number analyzed (Participants) | 41 | 36 | 45
days | 37 [29 to 57] | 43 [29 to 52] | 36 [29 to 50]

4. Secondary Outcome: Time to Stable Culture Conversion on Liquid MGIT Media
Description: Time (in days) to stable culture conversion on liquid MGIT media
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | RPT450 | RIF 600 | RPT 600
Number analyzed (Participants) | 31 | 46 | 45
days | 50 [38 to 61] | 59 [36 to 63] | 57 [43 to 62]

5. Secondary Outcome: Pharmacokinetics of Rifapentine
Description: area under the concentration time curve (AUC[0-24]) for rifapentine administered once daily at doses of 450 mg or 600 mg in the context of multi drug intensive phase TB treatment
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: ug x h/ml
Groups:
- Rifapentine 450 mg: Rifapentine 450 mg
- Rifapentine 600 mg: Rifapentine 600 mg
Arm/Group | Rifapentine 450 mg | Rifapentine 600 mg
Number analyzed (Participants) | 36 | 45
ug x h/ml | 330 [271 to 396] | 435 [294 to 504]

ADVERSE EVENTS:
Arm/Group | RPT450 | RIF 600 | RPT 600
Serious Adverse Events (participants affected / at risk) | 0/54 | 2/48 | 0/51
Other Adverse Events (participants affected / at risk) | 0/54 | 2/48 | 1/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RPT450 (N=54) | RIF 600 (N=48) | RPT 600 (N=51)
hospitalization (Infections and infestations) | 0 | 1 | 0 — hospitalization for lower respiratory tract infection
hospitalization for psychosis (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RPT450 (N=54) | RIF 600 (N=48) | RPT 600 (N=51)
hepatotoxicity (Hepatobiliary disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No